CLINICAL TRIAL: NCT01389596
Title: A DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP, MULTICENTER STUDY OF THE EFFICACY AND SAFETY OF PREGABALIN AS ADJUNCTIVE THERAPY IN CHILDREN 4 -16 YEARS OF AGE WITH PARTIAL ONSET SEIZURES
Brief Title: A Study of the Efficacy and Safety of Pregabalin as Add-On Therapy for Partial Onset Seizures in Children Ages 4-16 Years
Acronym: PERIWINKLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081041; 2010-020852-79 (EudraCT Number); XALCORY 1014 (Other: Alias Study Number)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2019-01

CONDITIONS: Epilepsy, Partial Seizures
Keywords: safety; efficacy; partial onset seizures; pediatric; pregabalin; placebo-controlled; double-blind
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Pregabalin add-on therapy
- Pregabalin Level 1 (max 150 mg/day) (Experimental)
  Interventions: Drug: Pregabalin add-on therapy
- Pregabalin Level 2 (max 600 mg day) (Experimental)
  Interventions: Drug: Pregabalin add-on therapy

INTERVENTIONS:
Drug: Pregabalin add-on therapy — Subjects will be randomized to receive a fixed dose of either placebo, pregabalin Level 1 (maximum 150 mg/day) or pregabalin Level 2 (maximum 600 mg/day) in a 1:1:1 ratio, in addition to the subjects current AED medication regimen. Either capsules or oral liquid form will be administered, depending on subjects preference and ability to swallow capsules, in two equally divided daily doses. The study will have an 8 week baseline period; a 2 week dose escalation period; a 9 week dose maintenance period; and a 1 week dose taper period.
  Arms: Placebo
Drug: Pregabalin add-on therapy — Subjects will be randomized to receive a fixed dose of either placebo, pregabalin Level 1 (maximum 150 mg/day) or pregabalin Level 2 (maximum 600 mg/day) in a 1:1:1 ratio, in addition to the subjects current AED medication regimen. Either capsules or oral liquid form will be administered, depending on subjects preference and ability to swallow capsules, in two equally divided daily doses. The study will have an 8 week baseline period; a 2 week dose escalation period; a 9 week dose maintenance period; and a 1 week dose taper period.
  Arms: Pregabalin Level 1 (max 150 mg/day)
Drug: Pregabalin add-on therapy — Subjects will be randomized to receive a fixed dose of either placebo, pregabalin Level 1 (maximum 150 mg/day) or pregabalin Level 2 (maximum 600 mg/day) in a 1:1:1 ratio, in addition to the subjects current AED medication regimen. Either capsules or oral liquid form will be administered, depending on subjects preference and ability to swallow capsules, in two equally divided daily doses. The study will have an 8 week baseline period; a 2 week dose escalation period; a 9 week dose maintenance period; and a 1 week dose taper period.
  Arms: Pregabalin Level 2 (max 600 mg day)

SUMMARY:
Study A0081041 is a double blind, placebo controlled, randomized, parallel group, multicenter study to evaluate the safety and efficacy of two dose levels of pregabalin administered in equally divided daily doses, in either capsule or oral liquid formulation, as adjunctive therapy in pediatric subjects 4 to 16 years of age with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or parent(s)/legally acceptable representative must be considered willing and able to sign consent, and complete daily seizure diaries and monitor seizure frequency.
* Male and female epilepsy subjects, 4 to 16 years of age inclusive on the date of the Screening Visit.
* Diagnosis of epilepsy with partial onset seizures classified as simple partial, complex partial or partial becoming secondarily generalized, according to the International League Against Epilepsy (ILAE) Diagnosis criteria.
* Must have a partial onset seizure frequency of at least 3 seizures per 28 day period prior to screening. Must have a partial onset seizure frequency of at least 6 seizures and no continuous 4 week seizure free period during the 8 week baseline phase prior to randomization.
* Currently receiving a stable dose of 1 to 3 antiepileptic drugs (stable within 28 days prior to screening).

Exclusion Criteria:

* Primary generalized seizures (including in the setting of co-existing partial onset seizures) which include, for example: Clonic, tonic and clonic-tonic seizures (note that partial onset seizures that become secondarily generalized are not exclusionary); Absence seizures; Infantile spasms; Myoclonic, myoclonic atonic, myoclonic tonic seizures.
* Lennox Gastaut syndrome, Benign Epilepsy with Centrotemporal Spikes (BECTS) and Dravet syndrome.
* A current diagnosis of febrile seizures, or seizures related to an ongoing acute medical illness. Any febrile seizures within 1 year of screening.
* Status epilepticus within 1 year prior to screening.
* Seizures related to drugs, alcohol, or acute medical illness.
* Any change in AED regimen (type of medication or dose) within 28 days of the Screening Visit or during the Baseline Phase.
* Progressive structural CNS lesion or a progressive encephalopathy.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 295 (Actual)
Dates: Start 2011-09-27 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (86):
- United States (20):
  - Center for Neurosciences, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children´s Hospital Los Angeles, Los Angeles, California
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Laszlo J. Mate, M.D., P.A., North Palm Beach, Florida
  - Pediatric Neurology, P.A., Orlando, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Center for Clinical and Translational Science, Lexington, Kentucky
  - Kentucky Neuroscience Institute, Lexington, Kentucky
  - University of Kentucky Hospital Epilepsy Monitoring Unit, Lexington, Kentucky
  - University of Kentucky Hospital Pharmacy, UK Chandler Hosptial, Lexington, Kentucky
  - Kosair Charities Pediatric Clinical, Louisville, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville Physicians, Louisville, Kentucky
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Duke Clinical Research Unit, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Road Runner Research, Ltd., San Antonio, Texas
- Belgium (3):
  - Centre Hospitalier Neurologique William Lennox, Ottignies, Brabant Wallon
  - HUDERF, Brussels, Brussels Capital
  - Cliniques Universitaires de Bruxelles Hôpital Erasme, Brussels
- UMBAL Sveti Georgi, Klinika po pediatria i genetichni zabolyavania, Plovdiv, Bulgaria
- Czechia (2):
  - Fakultni nemocnice Brno - Detska nemocnice, Brno - Cerna Pole
  - Fakultni nemocnice v Motole, Prague
- France (4):
  - CHU Bordeaux - Hopital des Enfants, Bordeaux
  - Hôpital Mère Enfant, Bron
  - Hopital Raymond Poincare, Garches
  - Hopitaux Universitaires de Strasbourg - Hopital Hautepierre, Strasbourg
- Greece (2):
  - General Childrens Hospital of Athens P & A Kyriakou, Athens
  - General Children's Hospital Penteli, Athens
- Hungary (6):
  - Dr. Kenessey Albert Korhaz es Rendelointezet, Balassagyarmat
  - Szent Janos Korhaz es Eszak Budai Egyesitett Korhazak, Budapest
  - Semmelweis Egyetem, I. Sz. Gyermekgyogyaszati Klinika, Budapest
  - Heim Pal Gyermekkorhaz, Neurologiai Osztaly, Budapest
  - Magyarorszagi Reformatus Egyhaz Bethesda Gyermekkorhaz, Gyermekneurologia, Budapest
  - Pécsi Tudományegyetem Klinikai Központ, Pécs
- Bnai Zion Medical Center, Haifa, Israel
- Italy (4):
  - A.O.U. Ospedali Riuniti di Ancona Presidio Ospedaliero G. Salesi, Ancona
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino, IRCCS - Servizio di Farmacia, Pavia
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino, IRCCS, Pavia
- Malaysia (2):
  - Paediatric Department, Ipoh, Perak
  - Hospital Kuala Lumpur, Kuala Lumpur
- Philippines (7):
  - Cebu Doctors' University Hospital, Cebu City, CEBU
  - Center for Neurodiagnostic and Therapeutic Services, Sta Cruz, Manila
  - Capitol Medical Center Inc., Quezon City, National Capital Region
  - Cebu Doctors' University Hospital, Cebu City
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
  - Philippine Children's Medical Center, Quezon City
- Poland (5):
  - Klinika Neurologii Rozwojowej, Gdansk
  - NZOZ Centrum Neurologii Dzieciecej i Leczenia Padaczki, Kielce
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. sw. Ludwika w Krakowie, Krakow
  - Katedra i Klinika Neurologii Wieku Rozwojowego, Poznan
  - Oddzial Neurologii Dzieciecej, Dolnoslaski Szpital Specjalistyczny im.T. Marciniaka, Wroclaw
- Romania (5):
  - Spitalul clinic de copii Dr. Victor Gomoiu, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Al. Obregia", Bucharest
  - Spitalul Clinic de Urgente pentru Copii "Sf. Maria",, Iași
  - Spitalul de Psihiatrie Dr. Ghe. Preda, Sibiu
  - Centrul Medical Dr. Bacos Cosma, Timișoara
- Serbia (4):
  - Institute for Child and Youth Healthcare of Vojvodina, Novi Sad, Vojvodina
  - Mother and Child Healthcare Institute Dr Vukan Cupic, Belgrade
  - University Children's Hospital Belgrade, Belgrade
  - Clinical Center of Kragujevac, Kragujevac
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- South Korea (3):
  - Samsung Medical Center/ Department of Pediatrics, Pediatric Neurology, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Turkey (Türkiye) (6):
  - Ege University Medical Faculty Department of Pediatrics Health and Diseases, Izmir, Bornova
  - Karadeniz Technical University Faculty of Medicine Farabi Hospital, Trabzon, Farabi
  - Izmir Tepecik Training and Research Hospital, Izmir, Konak
  - Behcet Uz Children Disease and surgery Training and research hospital, Izmir, Konak
  - Marmara University Pendik Training and Research Hospital, Istanbul, Pendik
  - Hacettepe University Medical Faculty, Ankara, Sihhiye/ankara
- Ukraine (9):
  - Komunalnyi zaklad "Dnipropetrovska dytiacha miska klinichna likarnia, Dnipropetrovsk
  - Komunalnyi zaklad "Dnipropetrovska oblasna dytiacha klinichna likarnia", Dnipropetrovsk
  - Derzhavna ustanova "Instytut nevrolohii, psykhiatrii ta narkolohii, Kharkiv
  - Derzhavna Ustanova Instytut Nevrolohii, Psykhiatrii ta Narkolohii NAMN Ukrainy,, Kharkiv
  - Derzhavnyi zaklad "Ukrainskyi medychnyi tsentr reabilitatsii ditei z, Kyiv
  - Komunalna ustanova "Odeskyi oblasnyi medychnyi tsentr psykhichnoho zdorovia",, Odesa
  - Komunalna ustanova "Odeska oblasna dytiacha klinichna likarnia", Oblasnyi tsentr rannoi, Odesa
  - Komunalna ustanova "Odeska oblasna psykhiatrychna likarnia 2",, S. Oleksandrivka
  - Oblasnyi klinichnyi tsentr neirokhirurhii ta nevrolohii, viddilennia neirokhirurhii 2,, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Antinew J, Pitrosky B, Knapp L, Almas M, Pitman V, Liu J, Craiu D, Modequillo M, Nordli D, Farkas V, Farkas MK. Pregabalin as Adjunctive Treatment for Focal Onset Seizures in Pediatric Patients: A Randomized Controlled Trial. J Child Neurol. 2019 Apr;34(5):248-255. doi: 10.1177/0883073818821035. Epub 2019 Jan 27. PMID 30688135
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081041&StudyName=A%20Study%20of%20the%20Efficacy%20and%20Safety%20of%20Pregabalin%20as%20Add-On%20Therapy%20for%20Partial%20Onset%20Seizures%20in%20Children%20Ages%204-16%20Years

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day: Participants aged 4 to 16 years and less than (<) 30 kilograms (kg) in weight, received pregabalin 3.5 milligram per kilogram per day (mg/kg/day) (up to a maximum of 150 mg/day) oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months). Participants aged 4 to 16 years and greater than or equal to (>=) 30 kg in weight, received pregabalin 2.5 mg/kg/day (up to a maximum of 150 mg/day) capsule or oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months).
- Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day: Participants aged 4 to 16 years and < 30 kg in weight, received pregabalin 14 mg/kg/day (up to a maximum of 600 mg/day) oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months). Participants aged 4 to 16 years and >= 30 kg in weight, received pregabalin 10 mg/kg/day (up to a maximum of 600 mg/day) capsule or oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months).
- Placebo: Participants aged 4 to 16 years received placebo matched to pregabalin, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months). Participants <30 kg in weight received placebo in the form of oral solution while participants >=30 kg in weight received placebo in the form of oral solution or capsule.
Period: Overall Study
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Started | 104 | 97 | 94
Completed | 94 | 81 | 84
Not Completed | 10 | 16 | 10
Not completed — Protocol Violation | 3 | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Insufficient Clinical Response | 3 | 4 | 5
Not completed — Adverse Event | 1 | 4 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Other Unspecified | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day: Participants aged 4 to 16 years and <30 kg in weight, received pregabalin 3.5 mg/kg/day (up to a maximum of 150 mg/day) oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months). Participants aged 4 to 16 years and >= 30 kg in weight, received pregabalin 2.5 mg/kg/day (up to a maximum of 150 mg/day) capsule or oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks (3 months).
- Total: Total of all reporting groups
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo | Total
Number analyzed (Participants) | 104 | 97 | 94 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (3.9) | 10.1 (3.5) | 10.3 (3.7) | 10.2 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 41 | 40 | 133
  Male | 52 | 56 | 54 | 162

OUTCOME MEASURES:

1. Primary Outcome: Log-Transformed 28-Day Seizure Rate For All Partial Onset Seizures During Baseline Phase
Description: All partial onset seizures experienced during baseline phase were recorded by the participants or their parents/legal guardian, in a daily seizure diary. 28-day seizure rate for all partial onset seizures = ([number of seizures in the baseline phase] divided by [number of days in baseline phase minus {-} number of missing diary days in baseline phase])*28. For log-transformation, the quantity 1 was added to the 28-day seizure rate for all participants to account for any possible "0" seizure incidence. This resulted in final calculation as: log transformed (28-day seizure rate +1).
Time Frame: Baseline phase (up to 8 weeks prior to treatment phase [Day 1])
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study drug during the double-blind treatment phase and had a baseline and at least 1 follow-up efficacy assessment.
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 93
Seizures per 28 days | 3.27 (1.215) | 3.19 (1.269) | 3.18 (1.302)

2. Primary Outcome: Log-Transformed 28-Day Seizure Rate For All Partial Onset Seizures During 12-Week Treatment Phase
Description: All partial onset seizures experienced during treatment phase were recorded by the participants or their parents/legal guardian in a daily seizure diary. 28-day seizure rate for all partial onset seizures = ([number of seizures in the treatment phase] divided by [number of days in treatment phase minus {-} number of missing diary days in treatment phase])*28. For log-transformation, the quantity 1 was added to the 28-day seizure rate for all participants to account for any possible "0" seizure incidence. This resulted in final calculation as: log transformed (28-day seizure rate +1).
Time Frame: Day 1 up to Week 12
Population: ITT population included all randomized participants who received at least 1 dose of study drug during the double-blind treatment phase and had a baseline and at least 1 follow-up efficacy assessment. Here, "Number of Participants Analyzed (N)" signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Seizures per 28 days
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 103 | 96 | 93
Seizures per 28 days | 2.86 (0.070) | 2.74 (0.072) | 2.96 (0.073)
Statistical Analysis 1: Comparison: Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day vs Placebo; Linear Model With Log transformed baseline seizure rate as continuous covariate and geographic regions, treatment groups and weight as fixed effects; Test type: Superiority or Other; p = 0.2577, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.29 to 0.08], Standard Error of Mean 0.092
Statistical Analysis 2: Comparison: Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0185, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.41 to -0.04], Standard Error of Mean 0.094

3. Secondary Outcome: Percentage of Participants With at Least 50 Percent (%) or Greater Reduction From Baseline in 28-day Seizure Rate During the 12 Week Treatment Phase
Description: Percentage of participants with 50 percent (%) or greater reduction from baseline in 28-day seizure rate during the 12 week treatment phase were reported. 28-day seizure rate for all partial onset seizures = ([number of seizures in the treatment phase] divided by [number of days in treatment phase minus {-} number of missing diary days in treatment phase])*28.
Time Frame: Day 1 up to Week 12
Population: ITT population included all randomized participants who received at least 1 dose of study drug during the double-blind treatment phase and had a baseline and at least 1 follow-up efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 93
percentage of participants | 29.1 | 40.6 | 22.6
Statistical Analysis 1: Comparison: Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day vs Placebo; P-values were from a Logistic Regression Model including fixed effects for treatment, weight group, and geographical region; Test type: Superiority or Other; p = 0.8024, Regression, Logistic; Odds Ratio (OR) = 1.036, 95% CI 2-sided [0.528 to 2.030]
Statistical Analysis 2: Comparison: Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0092, Regression, Logistic; Odds Ratio (OR) = 1.636, 95% CI 2-sided [0.851 to 3.147]

4. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 7 days after last dose of study drug (up to 13 weeks) that were absent before treatment or that worsened relative to pre- treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Day 1 up to 7 days after last dose of study drug (up to 13 weeks)
Population: Safety population included all randomized participants who took at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 94
participants
  AEs | 67 | 68 | 56
  SAEs | 5 | 10 | 7

5. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 7 days after last dose of study drug (up to 13 weeks) that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to drug was assessed by the investigator. AEs included both serious and non-serious adverse events.
Time Frame: Day 1 up to 7 days after last dose of study drug (up to 13 weeks)
Population: Safety population included all randomized participants who took at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 94
participants
  AEs | 37 | 46 | 30
  SAEs | 1 | 1 | 1

6. Other Pre Specified Outcome: Number of Adverse Events by Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs were classified according to the severity in 3 categories a) mild: AEs does not interfere with participant's usual function b) moderate: AEs interferes to some extent with participant's usual function c) severe: AEs interferes significantly with participant's usual function.
Time Frame: Day 1 up to 7 days after last dose of study drug (up to 13 weeks)
Population: Safety population included all randomized participants who took at least 1 dose of the study drug.
Measure: Number; unit: events
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 94
events
  Mild | 144 | 162 | 126
  Moderate | 33 | 31 | 21
  Severe | 7 | 3 | 5

7. Other Pre Specified Outcome: Number of Participants (6-16 Years of Age) With Positive Response to Columbia Suicide-Severity Rating Scale (C-SSRS) According to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories At Baseline
Description: The C-SSRS (mapped to C-CASA) is a participant-rated questionnaire to assess suicidal ideation and suicidal behavior. For suicidal ideation and behaviour, data from C-SSRS was mapped to C-CASA codes 1, 2, 3, 4 and 7. C-SSRS assessed whether participant experienced the following: completed suicide (C-CASA code 1); suicide attempt (response of "Yes" on "actual attempt") (C-CASA code 2); preparatory acts toward imminent suicidal behavior (ISB) ("Yes" on "preparatory acts or behavior")(C-CASA code 3); suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent) (C-CASA code 4); any self-injurious behavior with no suicidal intent (C-CASA code 7). In this outcome, number of participants with positive response (response of "yes") to C-SSRS (mapped to C-CASA categories 2, 3, 4 and 7) at baseline were reported.
Time Frame: Baseline (4 week prior to Day 1 of treatment)
Population: Safety population included all randomized participants who took at least 1 dose of the study drug. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 92 | 81 | 80
participants
  Suicide attempt (C-CASA code 2) | 0 | 0 | 0
  Preparatory acts towards ISB (C-CASA code 3) | 0 | 0 | 0
  Suicidal ideation (C-CASA code 4) | 0 | 0 | 0
  Self injurious behavior (C-CASA code 7) | 1 | 1 | 1

8. Other Pre Specified Outcome: Number of Participants (6-16 Years of Age) With Positive Response to Columbia Suicide-Severity Rating Scale (C-SSRS) According to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories During Post Baseline Time Period
Description: C-SSRS (mapped to C-CASA):participant-rated questionnaire to assess suicidal ideation and suicidal behavior. For suicidal ideation and behaviour, data from C-SSRS was mapped to C-CASA codes 1, 2, 3, 4 and 7. C-SSRS assessed whether participant experienced the following: completed suicide (C-CASA code 1); suicide attempt (response of "Yes" on "actual attempt") (C-CASA code 2); preparatory acts toward imminent suicidal behavior (ISB) ("Yes" on "preparatory acts or behavior")(C-CASA code 3); suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent) (C-CASA code 4); any self-injurious behavior with no suicidal intent (C-CASA code 7). Number of participants with positive response (response of "yes") to C-SSRS (mapped to C-CASA categories 1, 2, 3, 4 and 7) during post baseline time period (Day 1 up to Week 13) were reported
Time Frame: Day 1 up to Week 13
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 91 | 83 | 80
participants
  Completed suicide (C-CASA code 1) | 0 | 0 | 0
  Suicide attempt (C-CASA code 2) | 0 | 0 | 0
  Preparatory acts towards ISB (C-CASA code 3) | 0 | 0 | 0
  Suicidal ideation (C-CASA code 4) | 1 | 0 | 1
  Self injurious behavior (C-CASA code 7) | 1 | 2 | 2

9. Other Pre Specified Outcome: Child Behaviour Checklist (CBCL): Internalizing Subscale Score in Participants Less Than 6 Years of Age
Description: CBCL assessed suicidal behavior in children below 6 years. It is 100-item questionnaire completed by parent/legal guardian, based on participant's behavior in past 2 months. All 100 items rated on 3-point scale: 0=not true for that child; 1=sometimes true; 2=very/often true. Total CBCL score ranges from 0 (not true) to 200 (very/often true). Higher scores=higher levels of problematic behaviors or dysfunction. Scores from all items were used to calculate 3 subscale scores: Withdrawn subscale scores, Internalizing problems subscale scores and total problem subscale scores. All subscale scores reported scaled to T Scores. Higher scores for each CBCL subscales indicated higher levels of problematic behaviors or dysfunction. In this study, a cut-off of >=68 on the T-scores was used for all 3 subscales. If a participant T Score was >=68 in any of the sub-scales, the participant was referred for Mental Health Risk Assessment that included assessment of participant continuation to the study.
Time Frame: Week -8 (8 weeks prior to Day 1 of treatment), Week -4 (4 weeks prior to Day 1 of treatment), Day 1 (Week 0), Week 1, 2, 3, 6, 9, 12, end of study visit (Week 13)
Population: Safety population included all randomized participants who took at least 1 dose of the study drug.Here, "N" signifies number of participants who were evaluable for this measure and 'n' signifies number of participants evaluated for specific categories for each arm respectively.
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 12 | 14 | 14
T scores
  Week -8 (n= 12, 14, 14) | 48.3 (12.12) | 55.1 (9.37) | 54.9 (11.15)
  Week -4 (n= 12, 14, 14) | 48.1 (12.12) | 50.9 (7.01) | 52.6 (9.19)
  Week 0 (n= 12, 14, 14) | 46.4 (14.14) | 49.1 (7.08) | 50.6 (9.61)
  Week 1 (n= 12, 13, 14) | 46.3 (14.47) | 48.7 (9.36) | 50.7 (9.47)
  Week 2 (n= 11, 13, 13) | 46.5 (14.45) | 45.6 (8.21) | 48.3 (10.93)
  Week 3 (n= 12, 14, 13) | 45.6 (13.33) | 44.2 (9.37) | 49.6 (10.38)
  Week 6 (n= 11, 13, 11) | 45.5 (16.73) | 42.1 (9.65) | 47.5 (15.19)
  Week 9 (n= 11, 13, 11) | 46.0 (15.43) | 40.6 (10.19) | 51.0 (9.81)
  Week 12 (n= 11, 14, 13) | 42.1 (11.99) | 40.8 (8.95) | 50.5 (8.91)
  Week 13 (n= 12, 14, 11) | 44.3 (13.61) | 39.9 (7.77) | 50.8 (10.23)

10. Other Pre Specified Outcome: Child Behaviour Checklist (CBCL): Withdrawn Subscale Score in Participants Less Than 6 Years of Age
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 12 | 14 | 14
T scores
  Week -8 (n= 12, 14, 14) | 56.4 (6.04) | 64.0 (10.29) | 63.1 (10.50)
  Week -4 (n= 12, 14, 14) | 55.4 (5.43) | 61.3 (8.99) | 61.9 (10.48)
  Week 0 (n= 12, 14, 14) | 56.6 (6.68) | 60.6 (8.06) | 60.9 (10.86)
  Week 1 (n= 12, 13, 14) | 56.8 (7.12) | 60.9 (10.01) | 59.5 (10.09)
  Week 2 (n= 11, 13, 13) | 56.3 (6.17) | 60.2 (9.32) | 59.2 (11.61)
  Week 3 (n= 12, 14, 13) | 54.8 (6.80) | 58.6 (8.53) | 60.8 (11.02)
  Week 6 (n= 11, 13, 11) | 55.5 (8.29) | 56.6 (5.24) | 54.5 (20.82)
  Week 9 (n= 11, 13, 11) | 56.1 (6.99) | 57.1 (7.30) | 60.0 (10.64)
  Week 12 (n= 11, 14, 13) | 54.0 (5.48) | 57.3 (9.53) | 59.6 (10.11)
  Week 13 (n= 12, 14, 11) | 55.1 (6.43) | 56.1 (7.21) | 57.9 (10.58)

11. Other Pre Specified Outcome: Child Behaviour Checklist (CBCL): Total Problem Subscale Score in Participants Less Than 6 Years of Age
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 12 | 14 | 14
T scores
  Week -8 (n= 12, 14, 14) | 48.0 (10.84) | 50.7 (11.48) | 54.1 (10.94)
  Week -4 (n= 12, 14, 14) | 47.8 (11.04) | 47.0 (8.36) | 52.5 (7.35)
  Week 0 (n= 12, 14, 14) | 46.9 (11.75) | 45.2 (7.79) | 50.1 (8.81)
  Week 1 (n= 12, 13, 14) | 46.0 (13.65) | 43.8 (9.77) | 50.1 (8.40)
  Week 2 (n= 11, 13, 13) | 46.5 (13.17) | 42.1 (7.77) | 48.9 (8.95)
  Week 3 (n= 12, 14, 13) | 46.4 (12.64) | 42.4 (9.16) | 49.5 (9.81)
  Week 6 (n= 11, 13, 11) | 46.7 (15.25) | 38.7 (5.95) | 50.7 (8.86)
  Week 9 (n= 11, 13, 11) | 47.6 (13.13) | 38.4 (5.91) | 51.2 (9.12)
  Week 12 (n= 11, 14, 13) | 44.3 (11.78) | 39.0 (8.94) | 50.2 (9.28)
  Week 13 (n= 12, 14, 11) | 45.5 (13.28) | 37.9 (8.45) | 51.6 (9.53)

12. Other Pre Specified Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Scores at Week 12: Detection Task
Description: CogState battery:computerized test battery used to assess cognitive domains through cognition tests/tasks. The test battery was presented on computer with external response buttons. In this study, Cogstate battery consisted of 2 tasks which measured psychomotor function (detection task) and attention (paediatric identification task). Detection task was a measure of simple reaction time and provided a valid assessment of psychomotor function in participants. In this task, a playing card turning face up was presented in the center of the computer screen. As soon as this happened, the participant was to press the 'Yes' response key. There was no minimum or maximum scores since it was a time-based assessment. The software measured the speed of accurate responses to each event. In this outcome measure, speed of performance of participants (calculated as mean of the logarithmic base 10 transformed reaction times) for correct responses was reported. Lower scores indicated better performance.
Time Frame: Baseline (pre-dose at Day 1), Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: log10 milliseconds
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 74 | 61 | 66
log10 milliseconds
  Baseline (n= 68, 56, 60) | 2.71 (0.21) | 2.72 (0.20) | 2.70 (0.18)
  Change At Week 12 (n= 61, 45, 53) | -0.00 (0.12) | -0.03 (0.12) | 0.01 (0.09)

13. Other Pre Specified Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Week 12: Paediatric Identification (Go-No Go: Attention) Tasks
Description: CogState battery: computerized test battery used to assess cognitive domains through cognition tests/tasks. The test battery was presented on computer with external response buttons. Paediatric identification task: a measure of choice reaction time and valid assessment of visual attention. In this task, a playing card turning face up was presented in center of the computer screen. As soon as this happened, participant had to decide whether color of card was black or not. If color was black, participants was to press "Yes" response key, otherwise "no". There was no minimum/maximum scores since it was a time-based assessment. The software measured speed of accurate responses (correct identification of color) to each event. In this outcome measure, speed of performance of participants to correctly identify the color (calculated as mean of the logarithmic base 10 transformed reaction times) for correct responses was reported. Lower scores indicated better performance.
Time Frame: Baseline (pre-dose at Day 1), Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: log10 milliseconds
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 74 | 61 | 66
log10 milliseconds
  Baseline (n= 67, 56, 59) | 2.81 (0.15) | 2.80 (0.15) | 2.80 (0.14)
  Change At Week 12 (n= 60, 44, 51) | 0.00 (0.11) | 0.00 (0.12) | 0.00 (0.10)

14. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for abnormality: hematology (hemoglobin, hematocrit, red blood cells count:<]0.8*lower limit of normal [LLN],platelets:<0.5*LLN/greater than [>]1.75*upper limit of normal [ULN],leukocytes:<0.6*LLN or>1.5*ULN, lymphocytes, total neutrophils:<0.8*LLN or >1.2*ULN, basophils, eosinophil, monocytes:>1.2*ULN); Liver Function(aspartate aminotransferase ,alanine aminotransferase, alkaline phosphatase, Gamma glutamyl transferase:>0.3*ULN, total protein, albumin:<0.8*LLN or >1.2*ULN); bilirubin:>1.5*ULN; renal function(blood urea nitrogen, creatinine:>1.3*ULN); Electrolytes(sodium:<0.95*LLN or>1.05*ULN, potassium, chloride, calcium, bicarbonate:<0.9*LLN or >1.1*ULN); Lipids(cholesterol, triglycerides >1.3*ULN); creatine kinase:>2.0*ULN; glucose fasting:<0.6*LLN or >1.5*ULN, urine white blood corpuscles and RBC:>= 20/High Power Field [HPF];urine casts: >1/Low Power Field(LPF);urine bacteria:>20/HPF. Hormones (tetraiodothyronine and thyroid stimulating hormone:<0.8*LLN or >1.2*ULN).
Time Frame: Baseline (from 8 weeks prior to Day 1 of treatment) up to Week 13
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 102 | 95 | 93
participants | 61 | 63 | 61

15. Other Pre Specified Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for abnormalities in vital signs included: sitting systolic blood pressure (SBP) values: maximum increase and decrease of >=30 millimeter of mercury (mmHg) from baseline; sitting diastolic blood pressure (DBP) value: maximum increase and decrease of >=20 mmHg from baseline.
Time Frame: Baseline (from 8 weeks prior to Day 1 of treatment) up to Week 13
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 98 | 93 | 92
participants
  Maximum Increase from Baseline in Sitting SBP | 2 | 1 | 1
  Maximum Increase from Baseline in Sitting DBP | 6 | 8 | 11
  Maximum Decrease from Baseline in Sitting SBP | 5 | 1 | 1
  Maximum Decrease from Baseline in Sitting DBP | 15 | 6 | 10

16. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Neurological Examinations
Description: Neurological examinations included: level of consciousness, mental status, cranial nerve assessment, muscle strength and tone, reflexes, pin prick and vibratory sensation (the latter using a 128-Hertz tuning fork), coordination and gait. Clinical significance was based on investigator's discretion.
Time Frame: Baseline (from 8 weeks prior to Day 1 of treatment) up to Week 13
Population: Safety population included all randomized participants who took at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 94
participants | 0 | 1 | 0

17. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for abnormalities in ECG findings: 1) Time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS complex): >=140 milliseconds (msec); 2) The interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval): >=200 msec; 3) Time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula (QTCF interval): absolute value 450 to <480 msec, 480 to <500 msec, >=500 msec; 4) Maximum QT interval: >=500 msec; 5) Maximum QTCB interval (Bazett's correction): 450 to< 480 msec, 480 to <500 msec, >=500 msec. Only those categories of ECG abnormalities in which participants were found abnormal, were reported in this outcome measure.
Time Frame: Baseline (from 8 weeks prior to Day 1 of treatment) up to Week 13
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 102 | 97 | 94
participants
  Maximum PR Interval | 1 | 0 | 1
  Maximum QTCB Interval (Bazett's Correction) | 2 | 0 | 2

18. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examinations at Week 13
Description: Physical examinations evaluated the following body systems/organs: general appearance; dermatological; head and eyes; ears, nose, mouth, and throat; pulmonary; cardiovascular; abdominal; genitourinary (optional); lymphatic; musculoskeletal/extremities; and neurological. Clinical significance was determined by the investigator.
Time Frame: Baseline (from 8 weeks prior to Day 1 of treatment) up to Week 13
Population: Safety population included all randomized participants who took at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Number analyzed (Participants) | 104 | 97 | 94
participants | 5 | 5 | 2

ADVERSE EVENTS:
Arm/Group | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 5/104 | 10/97 | 7/94
Other Adverse Events (participants affected / at risk) | 66/104 | 64/97 | 55/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day (N=104) | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day (N=97) | Placebo (N=94)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Drug withdrawal convulsions (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 3 | 3
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin graft (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin: 2.5 mg/kg/Day or 3.5 mg/kg/Day (N=104) | Pregabalin: 10 mg/kg/Day or 14 mg/kg/Day (N=97) | Placebo (N=94)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 1
Myopia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Visual brightness (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 3 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 4 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Tooth erosion (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 4 | 4
Asthenia (General disorders) | 1 | 3 | 2
Energy increased (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 3
Feeling abnormal (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 9 | 9 | 7
Sluggishness (General disorders) | 0 | 2 | 0
Ascariasis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 3
Conjunctivitis (Infections and infestations) | 1 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Dermatitis infected (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 7 | 6
Otitis media (Infections and infestations) | 0 | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 3 | 2
Pharyngotonsillitis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 8 | 9
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 2 | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Ear abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2 | 3
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Gamma-glutamyl transferase increased (Investigations) | 1 | 0 | 1
Heart rate decreased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 4 | 13 | 4
White blood cell count increased (Investigations) | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 7 | 10 | 4
Overweight (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Clonus (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 3 | 1
Headache (Nervous system disorders) | 4 | 7 | 6
Hypersomnia (Nervous system disorders) | 2 | 1 | 2
Lethargy (Nervous system disorders) | 2 | 2 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 1 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 6 | 1 | 4
Somnolence (Nervous system disorders) | 18 | 25 | 13
Tunnel vision (Nervous system disorders) | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0
Disinhibition (Psychiatric disorders) | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 3 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 1
Mutism (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Tic (Psychiatric disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results